CLINICAL TRIAL: NCT00843713
Title: A Randomized, Controlled Trial Assessing the Effects of Raltegravir Intensification on Endothelial Function in Treated HIV Infection
Brief Title: Effect of Raltegravir on Endothelial Function in HIV-Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Priscilla Hsue, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01HL095130-01 (NIH)
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: HIV Infection; Inflammation; Cardiovascular Disease; HIV Infections
Keywords: HIV; endothelium; inflammation; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Inflammation; Cardiovascular Diseases | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): For subjects assigned to the placebo group, patients will take a matching placebo pill of 400 mg by mouth twice daily for 24 weeks in addition to taking their current HIV medication
  Interventions: Drug: Placebo
- Raltegravir (Active Comparator): For subjects assigned to the active comparator group, they will receive raltegravir at 400 mg by mouth twice daily for 24 weeks in addition to continuing to take their current HIV medication
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: raltegravir — For patients assigned to the raltegravir group, subjects will receive raltegravir 400mg to be taken by mouth twice daily for 24 weeks in addition to taking their current HIV medication
  Arms: Raltegravir
Drug: Placebo — For the patient assigned to the placebo group, subjects will take a matching placebo pill 400mg to be taken by mouth twice daily for 24 weeks in addition to taking their current HIV medication
  Arms: Placebo

SUMMARY:
Recent studies suggest that HIV patients are at increased risk for cardiovascular events; however, the mechanisms underlying this increased risk remain unclear. Our group was one of the first to demonstrate that HIV infection is independently associated with accelerated atherosclerosis, as measured by carotid artery-intima media thickness (IMT), and that HIV-associated inflammation may be driving this accelerated atherosclerosis. The mechanism by which HIV disease independent of any drug-specific toxicity increases the risk of cardiovascular disease during HAART is not known. We hypothesize that even well controlled HIV infection is independently associated with cardiovascular risk and that further decreasing HIV-associated inflammation adding newer antiretroviral agents will also decrease cardiovascular risk.

We will perform a small clinical trial of approximately 50 HIV-infected patients each to study the relationship between HIV infection, inflammation, thrombosis, atherogenic lipoproteins, and measures of atherosclerosis. We propose the following specific aims: Aim 1: To determine the influence of traditional and novel markers of inflammation on endothelial function and IMT progression; Aim 2: To determine if "intensification" with raltegravir in subjects on long-term antiretroviral therapy with clinically undetectable HIV RNA levels will improve endothelial function, and to determine if this effect is mediated by alterations in inflammatory markers, lipoproteins and/or thrombotic factors. For Aim 2, subjects from 2 randomized, double-blind, placebo-controlled raltegravir intensification studies will be asked to co-enroll in this cardiovascular study.

ELIGIBILITY:
Inclusion Criteria:

1. Stable antiretroviral therapy for at least 12 months
2. All plasma HIV RNA levels within the past year must be below level of detection (< 50 copies RNA/mL), although isolated single values > 50 but < 200 copies will be allowed.
3. Screening plasma HIV RNA levels < 50 copies RNA/mL
4. >90% adherence to therapy within the preceding 30 days, as determined by self-report
5. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
6. CD4<350 cells/mm3 for at least one year ("immunologic non-responder") or CD4>=350 cells/mm3 for at least one year ("immunologic responder").

Exclusion Criteria:

1. Ongoing or prior use of any integrase inhibitor or R5 inhibitor.
2. Patients who plan to modify existing antiretroviral therapy in the next 24 weeks for any reason
3. Serious illness requiring hospitalization or parental antibiotics within preceding 3 months
4. Concurrent or recent exposure to any immunomodulatory drugs
5. Advanced liver disease or active hepatitis B or C
6. Patients with systolic blood pressure <100/70
7. Starting or stopping statin therapy during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-01; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — San Francisco General Hospital
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Hatano H, Scherzer R, Wu Y, Harvill K, Maka K, Hoh R, Sinclair E, Palmer S, Martin JN, Busch MP, Deeks SG, Hsue PY. A randomized controlled trial assessing the effects of raltegravir intensification on endothelial function in treated HIV infection. J Acquir Immune Defic Syndr. 2012 Nov 1;61(3):317-25. doi: 10.1097/QAI.0b013e31826e7d0f. PMID 22918156

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Raltegravir
Started | 30 | 26
Completed | 30 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Raltegravir | Total
Number analyzed (Participants) | 30 | 26 | 56
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 53 [47 to 59] | 54 [47 to 59] | 53 [47 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 29 | 24 | 53
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 19 | 20 | 39
  African-American | 5 | 3 | 8
  Latino | 2 | 1 | 3
  Other | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function Measured by Brachial Artery Flow-mediated Dilation(FMD)
Description: Measurements in the change of brachial artery diameter from pre and post treatment.
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Placebo | Raltegravir
Number analyzed (Participants) | 30 | 26
millimeters | 3.4 [2.4 to 5.1] | 2.9 [2.6 to 5.1]

ADVERSE EVENTS:
Arm/Group | Placebo | Raltegravir
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/26
Other Adverse Events (participants affected / at risk) | 0/30 | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Raltegravir (N=26)
Hepatocellular Carcinoma (Hepatobiliary disorders) | 0 | 1 — The study MD does not believe this adverse event is related to study participation or study drug. Raltegravir has not been commonly associated with renal insufficiency.
Infection (Infections and infestations) | 1 | 0 — The principal investigator and co-principal investigator do not believe this adverse event was related to study participation. In addition to HIV, the subject has diabetes mellitus which may have predisposed him to getting the spinal infection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Raltegravir (N=26)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No